CLINICAL TRIAL: NCT02165891
Title: Prospective Randomized Study Comparing the Efficacy and Safety of Pleural Drainage by Video-Assisted Thoracoscopic With Pleural Drainage by Percutaneous Drain Associated With Urokinase in the Treatment of Parapneumonic Pleural Effusion in Children
Brief Title: Comparison of Intrapleural Urokinase and Video-Assisted Thorascopic Surgery in the Treatment of Parapneumonic Pleural Effusion in Children
Acronym: UROVATS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2013/PE1
Record Dates: First submitted 2014-02-26; First posted 2014-06-18 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Empyema, Pleural
MeSH Terms: conditions — Empyema, Pleural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urokinase (Other): insertion of a chest drain with urokinase instillation
  Interventions: Drug: insertion of a chest drain with urokinase instillation
- VATS (Other): primary video-assisted thorascopic surgery Other interventions except drainage procedure are the same in both arms
  Interventions: Procedure: primary video-assisted thorascopic surgery

INTERVENTIONS:
Drug: insertion of a chest drain with urokinase instillation — Other interventions except drainage procedure are the same in both arms
  Arms: Urokinase
Procedure: primary video-assisted thorascopic surgery
  Arms: VATS

SUMMARY:
Despite the improvement in the technology available for diagnosing and treating empyema, the management of empyema in children remains controversial.

The purpose of this study is to compare the efficacy and safety of two common technical approach used for pleural effusion drainage in the treatment of childhood empyema.

ELIGIBILITY:
Inclusion Criteria:

* patients under the age of 17
* pleural fluid depth of at least 15mm, confirmed by ultrasound
* at least one of the following severity criteria :

  1. fever continuing 48h after starting correct antibiotherapy
  2. respiratory distress
  3. mediastinal displacement on the chest X-ray

Exclusion Criteria:

* previous drainage by either Video-Assisted Thoracoscopic or pleural drainage by percutaneous drain associated with urokinase- congenital pulmonary disorders with lung function impairment
* congenital pulmonary disorders with lung function impairment
* chronic pulmonary disease associated with lung function impairment
* hemodynamic instability
* congenital immunodeficiency disease
* secondary immune deficiency induced
* hemostasis disorder (contraindication of thrombolytic therapy)
* pregnancy or breastfeeding patient

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
duration of drainage | end of drainage defined per protocole as < 1ml/kg/24h with an expected average time of two days to seven days

SECONDARY OUTCOMES:
length of hospital stay | Hospital departure with an expected average time of two weeks to one month
Duration of oxygen therapy | up to the end of patient hospitalisation with an expected average time of 48 hours to five days
duration of intravenous antibiotic therapy | up to the last intravenous antibiotic injection, minimum of 48 hours for a simple pleural effusion and a minimum of 14 days for an empyema with a maximum of one month
Duration of fever > 38.5°C | Up to fever resolution, with an average expected time of five days to 14 days
Number of Participants with Serious and Non-Serious Adverse Events | Up to the end of the hospitalisation, until three months corresponding to the end of follow up period
Patient discomfort | Up to chest drain removal with an average expected time of 48 hours up to seven days

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Fabiola University Children Hospital, Brussels, Belgium